CLINICAL TRIAL: NCT02509299
Title: Effect of Different Physiotherapy Treatments in Hospitalized COPD Patients
Brief Title: Effect of Physiotherapy in Hospitalized COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0055UG
Record Dates: First submitted 2015-07-19; First posted 2015-07-28 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: COPD
Keywords: COPD; NEMS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): patients will be involved in the Physiotherapy program 1. The program included 15 minutes of deep breathing exercises and 20-30 minutes of limb exercises. The exercises included global active range of motion (ROM) exercises and muscle strengthening like upper and lower limbs flexion-extension do single-leg stance, and sit to stand exercises added to standard treatment.
  Interventions: Other: Physiotherapy program 1
- Experimental group 2 (Experimental): patients will be involved in the physiotherapy program 2. The program was a combined intervention including the Control Group treatment plus neuromuscular stimulation therapy on quadriceps accompanied by lower limb exercises.
  Interventions: Other: Physiotherapy program 2
- Control group (Other): patients will receive standard medical treatment without physiotherapy intervention.
  Interventions: Drug: Standard medical treatment

INTERVENTIONS:
Other: Physiotherapy program 1 — The standard medical treatment and additionally they will receive physiotherapy. The program will be performed every day during the hospital stay and it will include global active range of motion (ROM) exercises and muscle strengthening like upper and lower limbs flexion-extension do single-leg stance, and sit to stand exercises.
  Other Names: Global exercises
  Arms: Experimental group 1
Other: Physiotherapy program 2 — COPD patients included in this group will receive the standard medical treatment and additionally, they will receive a physiotherapy program. The program will be performed every day during the hospital stay and included neuromuscular stimulation therapy on quadriceps accompanied by lower limbs exercises
  Other Names: NEMS and lower limb exercises
  Arms: Experimental group 2
Drug: Standard medical treatment — The standard medical treatment consists on:
  * Inhaled bronchodilators: Short acting inhaled β2 agonists ( salbutamol and terbutaline) and anticholinergic agents (ipratropium and oxitropium bromide).
  * Glucocorticoids:
  Inhaled glucocorticoids including beclomethasone dipropionate, budesonide, flunisolide, fluticasone propionate and triamcinolone acetonide, depending on the expert criteria.
  - Antibiotics: The antibiotics were administered according to the GOLD criteria including the β-lactamase inhibitor and fluoroquinolones.
  Other Names: Drugs
  Arms: Control group

SUMMARY:
Chronic obstructive pulmonary disease (COPD) impacts negatively on the balance and strength of patients. Several studies have shown that acute exacerbations (AEs) decrease, pulmonary function and survival of COPD patients, and there are a lot of physiotherapy interventions to improve it during the hospital stay.

The objective of the present study is to examine the effects of a physical therapy program on balance and strength in COPD patients hospitalized due to acute exacerbation.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major cause of morbidity and mortality worldwide. It is a progressive disease, characterized by lung function impairment with airway obstruction.

Patients with COPD suffer exacerbations; the frequency of these exacerbations increases with the severity of the disease. It has been previously shown that the level of health-related quality of life of COPD subjects deteriorates considerably with increasing severity of disease and that the deterioration is linearly related to a decrease in FEV1 % predicted normal values.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis with exacerbation.
* No contraindication of physiotherapy.
* Signed written consent.
* Medical approval for inclusion.

Exclusion Criteria:

* Contraindications for physiotherapy
* Neurological, orthopedic or heart disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
Lower limb strength | Participants will be followed for the duration of hospital stay, an expected average of 9 days.
  Lower limb strength was evaluated by a dynamometer. The assessor placed the limb to be examined in the starting position (a knee flexion of 90º) and instructed each participant to hold the limb in that position against the increasing resistance applied to it by the examiner. During each test the assessor counted out loud for seconds and at the end of the test period advised the participant to relax the limb.
Balance | Participants will be followed for the duration of hospital stay, an expected average of 9 days.
  Balance was evaluated by the one-leg standing balance test, that measured the time that the patient balance on one leg as long as possible. We asked the subject being tested to choose a leg to stand on (whichever he felt more comfortable with), flex the opposite knee allowing the foot to clear the floor, and balance on one leg as long as possible

SECONDARY OUTCOMES:
Respiratory function | Participants will be followed for the duration of hospital stay, an expected average of 9 days.
  Spirometry is regarded as the gold standard measure of respiratory function. The indicators of forced vital capacity (FVC) and forced expiratory volume in one second (FEV1) will be tested. Spirometry will be performed according to American Thoracic Society (ATS) criteria.
Anxiety and depression | Participants will be followed for the duration of hospital stay, an expected average of 9 days.
  The hospital anxiety and depression scale (HADS) will be used to evaluate psychological status. HADS is a 14-items self-report questionnaire designed to detect psychological morbidity in medically ill patients. It contains depression and anxiety subscales, each with scores ranging from 0 to 21.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Department of Physical Therapy, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided